CLINICAL TRIAL: NCT03694223
Title: A Feasibility Study on Different Health Education Delivery Methods for a Low Fermentable Carbohydrate (FODMAP) Diet in Patients With Functional Bowel Disorders
Brief Title: Health Education Delivery Methods for a Low Fermentable Carbohydrate Diet in Patients With Functional Bowel Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 206464
Record Dates: First submitted 2018-07-23; First posted 2018-10-03 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-07

CONDITIONS: Irritable Bowel Syndrome; Functional Diarrhea; Functional Bowel Disorder
Keywords: FODMAP; DIET; BLOATING
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Booklets (Experimental): Health education delivery method: Booklet. Patients will be given 2 leaflets on the low FOMDAP diet produced by the Department of Nutrition and Dietetic in Guy's & St Thomas' NHS Foundation Trust, and the Diabetes and Nutritional Sciences Division at King's College London. These booklets have been produced by dietitians and are commonly used in clinical practice across the UK.
  Interventions: Other: Health education delivery methods
- Mobile application (Experimental): Health education delivery method: Mobile application. Patients will be asked to download an application on their mobile phones or tablets. This application has been produced by dietitians from the Department of Nutrition and Dietetic in Guy's & St Thomas' NHS Foundation Trust, and the Diabetes and Nutritional Sciences Division at King's College London.
  Interventions: Other: Health education delivery methods
- One to one consultation with dietitian (Active Comparator): Health education delivery method:One-to-one consultation with dietitian. Patients will attend a clinic visit for a one-to-one consultation with a dietitian. As per current clinical practice, the initial visit will last for 1 hour. During the visit, tailored information on the low FOMDAP diet will be given to match patients' individual needs. During the visit, either the leaflets (used in group 1) or the application (used in group 2) will be used to facilitate the visit. The choice of using the leaflets or the app during the visit will be based on the dietitian's judgment based on the patients' needs.
  Interventions: Other: Health education delivery methods

INTERVENTIONS:
Other: Health education delivery methods

SUMMARY:
There is evidence for the use of a diet low in short chain fermentable carbohydrates (low FODMAP diet) in the management of functional gut symptoms, such as abdominal pain and bloating. However, the provision of advice on the low FODMAP diet can be challenging due to limited resources and the need for a dietitian with expertise in the low FODMAP diet. The aim of this study is to assess the feasibility in terms of recruitment and retention in planning a future trial. The purpose of the future trial will be to investigate the clinical and cost effectiveness, as well as the acceptability of different education methods of the low FODMAP diet for the treatment of IBS.

To date, there are no studies on the implementation of the low FOMDAP diet using a mobile app or leaflets in the education of the low FODMAP diet. Therefore, a feasibility study design was chosen in order to obtain key data on recruitment and retention rates at each study group.

DETAILED DESCRIPTION:
A low FODMAP diet includes FODMAP restriction, FODMAP re-introduction and FODMAP personalisation. This study will focus on FODMAP restriction whereby foods high in FODMAPs are avoided for 4 weeks.

Patients with IBS will be recruited from primary and secondary care centres.

STUDY GROUPS

Group 1: 2 x Booklets produced produced by the Department of Nutrition and Dietetic in Guy's & St Thomas' NHS Foundation Trust, and the Diabetes and Nutritional Sciences Division at King's College London. These booklets have been produced by dietitians and are commonly used in clinical practice across the UK. They contain the following information:

Group 2: Patients will be asked to download an application on their mobile phones or tablets. This application has been produced by dietitians from the Department of Nutrition and Dietetic in Guy's & St Thomas' NHS Foundation Trust, and the Diabetes and Nutritional Sciences Division at King's College London.

Group 3:Patients will attend a clinic visit for a one-to-one consultation with a dietitian. As per current clinical practice, the initial visit will last for 1 hour.

PRIMARY OBJECTIVE The primary objective is to estimate recruitment and retention rates of patients with IBS receiving different education delivery methods of the low FODMAP diet.

SAMPLE SIZE As this is a feasibility study, a formal sample size calculation is not appropriate. For such feasibility studies, sample sizes between 24 and 50 have been recommended. Therefore, for this study, a total sample size of 45 was chosen (15 patients per group). Previous work indicates an approximately 12% attrition rate and, therefore, the final sample size will be 50 patients.

ANALYSIS Descriptive statistics such as mean values, standard deviations (SD) for continuous variables, and counts (percentages) and confidence intervals (CI) for categorical variables will be calculated. To assess recruitment and retention rates the following will be recorded: number of people directly contacting the researchers for the study, number of participants pre-screened and screened, number of participants randomised, number of drop-outs.

ETHICS AND REGULATORY APPROVALS The trial will be conducted in compliance with the principles of the Declaration of Helsinki (1996), the principles of Good Clinical Practice. Ethical approval for this study has been granted by an NRES Committee London.

DATA HANDLING

The Chief Investigator will act as custodian for the trial data. The following guidelines will be strictly adhered to:

1. Patient data will be anonymised
2. All trial data will be stored on a password protected computer and limited to authorised study personnel
3. All records and samples will be stored in a secure environment
4. All trial data will be stored in line with the Data Protection Act
5. Data and samples will be securely stored for 5 years after the study has ended and may be used for further in depth analysis
6. Data may be accessed by regulatory authorities for audit purposes

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 or over with IBS, functional diarrhoea or functional bloating based on Rome IV criteria who do not have a major medical condition (diabetes, psychiatric or current eating disorders), gastrointestinal disease (e.g. inflammatory bowel disease, coeliac disease) or history of previous GI surgery, except cholecystectomy and haemorrhoidectomy
2. Individuals with no adequate relief of their symptoms at baseline, as well as those with frequency of abdominal pain or discomfort for 1 or more days/week.
3. Individuals with a BMI of 18.5 kgm2 or more.
4. Individuals able to give informed consent
5. Individuals able to understand English
6. Individuals able to read English
7. Individuals with access to Internet
8. Individuals with smartphone with Android or IOS (Apple) software who are able to download apps.

Exclusion Criteria:

1. Females who report to be pregnant or lactating
2. Individuals with constipation predominant IBS (IBS-C) based on the Rome IV criteria
3. Consumption of antibiotics, in the last 4 weeks prior to the study
4. Individuals with additional specific dietary needs (based on the dietitian's judgment)
5. Individuals with multiple food allergies
6. Individuals who have participated in other trials with investigational products within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
RECRUITMENT RATE | Baseline visit (Day 0)
  Recruitment rate of patients receiving different education delivery methods of the low FODMAP diet.
RETENTION RATE (overall and within each study group) | Follow-up visit (week 4)
  Retention rate of patients receiving different education delivery methods of the low FODMAP diet.

SECONDARY OUTCOMES:
Compliance rates to the diet | Follow-up visit (week 4)
  Compliance rates to the diet within the study groups assessed via a 7day food and drink diary
Satisfaction over the education delivery methods received | Baseline (Day 0) and Follow-up visit (week 4)
  Satisfaction over the education methods and diet, assessed via 5-point Likert scales (1=Strongly Agree, 2=Agree, 3=Neutral, 4=Disagree, 5=Strongly Disagree)
Appropriateness of the education methods received in each study group | Baseline (Day 0) and Follow-up visit (week 4)
  Perceived appropriateness of the education methods, assessed via 5-point Likert scales (1=Strongly Agree, 2=Agree, 3=Neutral, 4=Disagree, 5=Strongly Disagree)
Perceived fit of the education delivery methods within the NHS | Follow-up visit (week 4)
  Assessed via a 5-point Likert scale (1=Strongly Agree, 2=Agree, 3=Neutral, 4=Disagree, 5=Strongly Disagree)
Willingness of participants being assigned to the study groups using a multiple choice questionnaire. | Follow-up visit (week 4)
  Assessed via a question on whether they would like to have been randomised to a different group (Yes/No)
Gastrointestinal symptom severity | Baseline (Day 0) and Follow-up visit (week 4)
  Validated Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) questionnaire. The questionnaire includes four VAS items evaluating abdominal pain frequency and intensity, abdominal distension, satisfaction with bowel habit, and quality of life. Scores are then added up; scoring allows categorisation of patients into mild (75-174), moderate (175-300) and severe (>300) cases, with a maximum achievable severity score of 500 points. A minimal clinically important difference of a 50-point reduction in score allows meaningful interpretation of score change over time.
Health-related quality of life in irritable bowel syndrome | Baseline (Day 0) and Follow-up visit (week 4)
  Validated Irritable Bowel Syndrome-Quality of Life (IBS-QoL) questionnaire. Each item utilises a 5-point Likert response scale, which is transformed to a 0-100 point scale and subscale scores are then calculated (dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, relationships). A total score can be calculated by summing the subscale scores. A score of 100 denotes maximum QOL for subscales and the total score.
Gastrointestinal symptoms experienced | Baseline and follow-up visitBaseline (Day 0) and Follow-up visit (week 4)
  Assessed using Gastrointestinal Symptom Rating Scale (GSRS). Gastrointestinal symptoms (Abdominal discomfort or pain, Heartburn, Acid reflux, nausea, abdominal gurgling, bloating, burping, flatulence, constipation, diarrhoea, loos stools, hard stools, urgency, incomplete evacuation, tiredness, overall symptoms) are rated in a 4-point Likert scale (0=Absent, 1=Mild, 2=Moderate, 3=Severe). Descriptive and inferential statistical results are presented for each individual symptom seperately.
Adequate relief of symptoms | Baseline (Day 0) and Follow-up visit (week 4)
  Assessed using the "adequate relief of IBS symptoms" question (IBS-AR). The outcome is dischotomous (Yes/No) and counts/percentages that have reported adequate relief ("Yes") will be presented.
Estimates of the parameters required for calculation of the sample size for a future larger study | Screening (Week -1), Baseline (Day 0) and Follow-up visit (week 4)
  The results of this study will be used to inform the sample size calculation of a future larger study if needed. The outcome that will be used for the sample size calculation depends on the which the primary outcome of the future study will be. The mean and standard deviation generated from this study will be used for the sample size of the future trial.

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Lomer, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No